CLINICAL TRIAL: NCT02774551
Title: Physical Activity Intervention Trial to Mitigate Muscle Loss and Increase Muscle Strength in Esophageal Cancer Survivors
Brief Title: Physical Activity Intervention Trial to Mitigate Muscle Loss and Increase Muscle Strength
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed for recruitment March 2020 due to the ongoing covid-19 situation and the termination of the study inclusion was done in August 2020.
Sponsor: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA study
Record Dates: First submitted 2016-04-28; First posted 2016-05-17 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Oesophageal Cancer
Keywords: Body composition; Muscle strength; Health related quality of life
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity intervention group (Experimental): The physical activity program includes 150 minutes of minimum intensity activity during a week (e.g. walking, swimming) and five strength training exercises (10 repetitions and 2 sets of: squats, wall push ups, rowing with resistance band, shoulder press with resistance band, hip abduction) targeting the major muscle groups to do twice a week are demonstrated by the research nurse. The resistance training is progressive by increasing resistance in the band based on patient's adaptability during the intervention.
  Interventions: Behavioral: Physical activity intervention group
- Standard care control group (No Intervention): Patients follow their routine daily physical activity.

INTERVENTIONS:
Behavioral: Physical activity intervention group — 150 minutes of minimum intensity activity during a week (e.g. walking, swimming) and five strength training exercises (10 repetitions and 2 sets of: squats, wall push ups, rowing with resistance band, shoulder press with resistance band, hip abduction) targeting the major muscle groups to do twice a week.
  Arms: Physical activity intervention group

SUMMARY:
This intervention study will be conducted on patients included in a nationwide and prospective cohort, The Oesophageal Surgery in Cancer patients: Adaptation and Recovery study (OSCAR). The OSCAR includes patients operated on for oesophageal cancer in Sweden between 2013-2018, identified through pathology departments and included in the cohort 1 year after surgery. A comprehensive interview is conducted by a research nurse during a home visit using patient reported outcomes on several HRQOL, psychosocial, emotional and nutritional aspects. Regular follow-ups are carried out at 1½, 2, 2½, 3, 4 and 5 years postoperatively.

All patients within OSCAR are invited to the intervention trial. Half of the eligible patients will be randomised to intervention and half to standard care (control group) by means of block randomisation method. The intervention group will be encouraged to adhere to a physical activity regimen of 150 minutes of weekly minimum intensity activities and 5 simple strength training exercises twice a week as instructed by the research nurse. The control group will follow their routine daily physical activity. HRQOL measures, height and weight, body composition, muscle strength, functional mobility and strength, and dietary intake are assessed before and after the intervention. Compliance will be ensured by means of a daily physical activity dairy and a weekly follow up on telephone with all patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients from the nationwide prospective cohort the Oesophageal Surgery in Cancer patients: Adaptation and Recovery study (OSCAR) with willingness to participate

Exclusion Criteria:

* Current malignancies or co-morbidities, psychological or social conditions that prevent participation
* Patients with pacemakers; cochlear or other electrical implants cannot be screened using the bio-impedance scale for safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related increase in muscle mass as assessed by a bio-impedance body composition scale. | At baseline and after the 12 weeks intervention/control programme.
  The main outcome measure will be increase in skeletal muscle mass using a bio-impedance analysis portable monitor. Changes occurring during the period just before and just after the 12-weeks intervention programme, or standard of care in the comparison group, will be compared between the intervention group.
Number of participants with treatment related increase in muscle strength as assessed by a hand grip dynamometer and chair stand test. | At baseline and after the 12 weeks intervention/control programme.
  The main outcome measure will be increase in skeletal muscle strength using a handgrip dynamometer and 30 second sit stand test. Changes occurring during the period just before and just after the 12-weeks intervention programme, or standard of care in the comparison group, will be compared between the intervention group.

SECONDARY OUTCOMES:
Number of participants with improvement in physical function scale of health related quality of life as assessed from the questionnaire - European Organization for Research and Treatment of Cancer (EORTC); Quality of Life Questionnaire (QLQ) - C30. | At baseline and after the12 weeks intervention/control programme.
  This secondary outcome will assess the physical function scale of HRQOL using EORTC QLQ-C30 questionnaires before and after the intervention.
Number of participants with improvement in fatigue scale of health related quality of life as assessed from the questionnaire - EORTC QLQ-FA13. | At baseline and after the12 weeks intervention/control programme.
  This secondary outcome will assess the fatigue scale of HRQOL using EORTC fatigue questionnaire QLQ-FA13 before and after the intervention.
Number of participants with improvement in appetite loss function of health related quality of life as assessed from the oesophageal disease specific module - EORTC QLQ-OG25. | At baseline and after the12 weeks intervention/control programme.
  This secondary outcome will assess the appetite loss function of HRQOL using EORTC QLQ-OG25 questionnaire before and after the intervention.
Number of participants with improvement in eating difficulties scale of health related quality of life as assessed from the cachexia module of EORTC - QLQ-CAX24. | At baseline and after the12 weeks intervention/control programme.
  This secondary outcome will assess the eating difficulties scale of HRQOL using EORTC QLQ-CAX24 questionnaire before and after the intervention.
Number of participants with improvement in psycho social issues as assessed from the questionnaire - Hospital Anxiety and Depression Scale (HADS). | At baseline and after the12 weeks intervention/control programme.
  This secondary outcome will assess the psychosocial issues using HADS questionnaire before and after the intervention.
Number of participants with improvement in physical activity level measured using the international physical activity questionnaire (IPAQ). | At baseline and after the 12 weeks intervention/control programme.
  This secondary outcome shall include changes in the total physical activity level measured using the international physical activity questionnaire (IPAQ) before and after the intervention.
Number of participants with improvement in dietary intake measured using 3 day food diary. | Just before (baseline) and just after (final follow up) the 12 weeks intervention programme.
  This secondary outcome shall include changes in dietary intake measured using food dairy measured thrice a week: two weekdays and 1 weekend day before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Lagergren, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Surgical cares sciences, Karolinksa Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anandavadivelan P, Malberg K, Vikstrom K, Nielsen S, Holdar U, Johar A, Lagergren P. Home-based physical activity after treatment for esophageal cancer-A randomized controlled trial. Cancer Med. 2023 Feb;12(3):3477-3487. doi: 10.1002/cam4.5131. Epub 2022 Aug 18. PMID 36812121